CLINICAL TRIAL: NCT00340509
Title: A Genome-Wide Scan For Quantitative Trait Loci of Serum Bilirubin - A Framingham Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902016; 02-H-N016
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2013-07-23

CONDITIONS: Genetics
Keywords: Genetics; Population; CHD Risk; Epidemiology; Gene Mapping

SUMMARY:
Studies have shown that there is a significant association between serum bilirubin concentrations and risk of coronary artery disease (CAD). So far, no linkage analysis in humans between serum bilirubin and DNA markers has been reported. The purpose of this protocol is to identify chromosome regions that contain quantitative trait loci (QTL) involved in serum bilirubin metabolism and bilirubin concentration. In the Framingham Study, a 10cM genome scan (about 400 markers) has been conducted in more than three hundred families. Serum bilirubin was measured in the first and second exams of the Framingham Offspring. These data provide us the opportunity to undertake linkage analyses to map QTL of serum bilirubin.

DETAILED DESCRIPTION:
Many studies showed that there is a significant relationship between serum bilirubin levels and risk of coronary artery disease (CAD). We carried out a genome-wide scan for quantitative trait loci of serum bilirubin through the 330 extended Framingham families and found significant evidence of linkage of serum bilirubin to chromosome 2q telomere where an important candidate gene, Uridine diphosphate glycosyltransferase 1 gene (UGT1A1), resides. The purposes of this protocol are to confirm linkage between serum bilirubin and UGT1A1, mathematical modeling and association studies between the genotypes of UGT1A1 and CAD.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study population will include the members of the 330 Framingham Study families and 1888 random individuals.

The Original Cohort will also be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1888 (Actual)
Dates: Start 2001-10-26; Study Completion 2013-07-23

CONTACTS AND LOCATIONS:
Overall Officials: Gang PH Zheng, Ph.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Djousse L, Levy D, Cupples LA, Evans JC, D'Agostino RB, Ellison RC. Total serum bilirubin and risk of cardiovascular disease in the Framingham offspring study. Am J Cardiol. 2001 May 15;87(10):1196-200; A4, 7. doi: 10.1016/s0002-9149(01)01494-1. No abstract available. PMID 11356398
- [Background] Breimer LH, Wannamethee G, Ebrahim S, Shaper AG. Serum bilirubin and risk of ischemic heart disease in middle-aged British men. Clin Chem. 1995 Oct;41(10):1504-8. PMID 7586525
- [Background] Almasy L, Blangero J. Multipoint quantitative-trait linkage analysis in general pedigrees. Am J Hum Genet. 1998 May;62(5):1198-211. doi: 10.1086/301844. PMID 9545414